CLINICAL TRIAL: NCT02758691
Title: Examining the Neural Correlates of Memory in Response to Intranasal Insulin Through fMRI & Device Testing
Brief Title: fMRI Study of Effects of Nasal Insulin on Memory
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Rosalyn Moran, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VT15-462
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Human Memory; Intranasal Insulin
Keywords: memory; insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal Insulin (Experimental): Healthy participants will self-administer 20 IU of Humulin® R U-100 with the Precision Olfactory Delivery (POD) delivery device and complete a memory task in an fMRI (functional Magnetic Resonance Imaging) scanner.
  Interventions: Drug: Intranasal Insulin
- Saline Placebo (Placebo Comparator): Healthy participants will self-administer a saline solution with the Precision Olfactory Delivery (POD) delivery device and complete a memory task in an fMRI (functional Magnetic Resonance Imaging) scanner.
  Interventions: Drug: Intranasal Saline

INTERVENTIONS:
Drug: Intranasal Insulin — All participants in the devise testing portion of the study will self-administer a 20 IU dose of intranasal insulin. Half of the participants in the function Magnetic Resonance Imaging portion of the study will also self-administer a 20 IU dose of intranasal insulin.
  Other Names: Humulin® R U-100
  Arms: Intranasal Insulin
Drug: Intranasal Saline — All participants in the devise testing portion of the study will self-administer a 20 mL dose of intranasal saline. Half of the participants in the function Magnetic Resonance Imaging portion of the study will also self-administer a 20 mL dose of intranasal saline.
  Other Names: Sterile Water
  Arms: Saline Placebo

SUMMARY:
Recent research has suggested insulin may be involved in how human's form and recall memories. This study is designed to look at how nasal insulin is used in the brain. Specifically, how insulin alters the various connections within brain regions that occur while adults perform simple attention and memory tasks. This study is divided into two parts: blood draw procedure and fMRI (functional Magnetic Resonance Imaging) procedure. The blood draw procedure is designed to look at the effects of intranasal insulin using a Precision Olfactory Delivery (POD) device on the blood levels of glucose and insulin. Those asked to participate will receiving a low-dose saline solution and low-dose of insulin through a nasal spray followed by a blood draw session to measure your blood glucose and insulin levels over a 90 minute period.

Participation in the fMRI (functional Magnetic Resonance Imaging) procedure will involve receiving a low-dose of insulin or a saline solution through a nasal spray using a Precision Olfactory Delivery (POD) device and brain scan using Magnetic Resonance Imaging (MRI). During the scan, participants will complete a series of memory tasks reflected on a computer screen. The trial will be randomized and double-blinded.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults over the age of 18

Exclusion Criteria:

* any existing health conditions: including diabetes, history of alcoholism or drug dependence
* contraindications to Magnetic Resonance Imaging (MRI): any non-titanium metal in the head or body

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Change in Memory Recall Performance during functional Magnetic Resonance Imaging task | 1 day
  Recall performance will be measured based off a forced recall memory task. Participants will be asked to categorizes images as indoor or outdoor during an encoding task and then show a series of images and asked to indicated if the pictures is 'old' or 'new' in a recall task. The score will be calculated as a percentage of images correctly identified as 'old.'